CLINICAL TRIAL: NCT00800930
Title: Therapeutic Induction of Endogenous Antibiotics for Improved Recovery in Shigellosis
Brief Title: Therapeutic Induction of Endogenous Antibiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2004-031
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Shigellosis
Keywords: Shigellosis; sodium butyrate; antimicrobial peptides; LL-37; innate immunity; The aims are to assess efficacy of sodium butyrate enema in; marked improvement in clinical features; endoscopic findings; histological features; Induction of LL-37 in the rectum.
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Butyric Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients will be instructed to lie on a bed (cholera cot) in left lateral position. A soft rectal catheter will be introduced by a nurse/physician, through which 80 ml of butyrate solution will be instilled slowly with a 50 ml plastic syringe. Patients will be asked to retain the enema for at least ½ hour by remaining supine for 30 minutes after the administration. However, if a patient cannot retain the enema for 30 minutes, he will be given a second round of enema immediately after defecation.
  Interventions: Biological: Sodium Butyrate
- 2 (Placebo Comparator): Patients will be instructed to lie on a bed (cholera cot) in left lateral position. A soft rectal catheter will be introduced by a nurse/physician, through which 80 ml of saline solution will be instilled slowly with a 50 ml plastic syringe. Patients will be asked to retain the enema for at least ½ hour by remaining supine for 30 minutes after the administration. However, if a patient cannot retain the enema for 30 minutes, he will be given a second round of enema immediately after defecation.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Sodium Butyrate — Patients will be instructed to lie on a bed (cholera cot) in left lateral position. A soft rectal catheter will be introduced by a nurse/physician, through which 80 ml of butyrate solution will be instilled slowly with a 50 ml plastic syringe. Patients will be asked to retain the enema for at least ½ hour by remaining supine for 30 minutes after the administration. However, if a patient cannot retain the enema for 30 minutes, he will be given a second round of enema immediately after defecation.
  Arms: 1
Biological: Saline — Patients will be instructed to lie on a bed (cholera cot) in left lateral position. A soft rectal catheter will be introduced by a nurse/physician, through which 80 ml of saline solution will be instilled slowly with a 50 ml plastic syringe. Patients will be asked to retain the enema for at least ½ hour by remaining supine for 30 minutes after the administration. However, if a patient cannot retain the enema for 30 minutes, he will be given a second round of enema immediately after defecation.
  Arms: 2

SUMMARY:
Shigellosis is one of the major causes of morbidity and mortality in many developing countries. The continued emergence of antibiotic resistant strains has complicated the treatment of shigellosis and has increased the cost of treatment markedly. Antimicrobial peptides are considered as endogenous antibiotic. A mixture of these antimicrobial peptides (LL-37 and beta-defensin) drenches the mucosal epithelial surfaces forming a barrier for invading microorganisms. Recently, we found that Shigella down-regulates the expression of LL-37 and beta-defensin 1 (HBD-1) in the colon of patients during acute shigellosis thereby facilitating bacterial invasion. Both LL-37 and HBD-1 could inhibit the growth of various microbes e.g. S. dysenteriae type 1, S. flexneri, and S. boydii. Our study indicated that bacterial DNA might be a potential mediator for the down- regulation in vitro. Down-regulation of LL-37 and HBD-1 was also seen in watery diarrhea caused by other pathogens. Thus, bacteria-mediated down-regulation of our front line defenses could be one strategy evolved by the pathogens to subvert this host-defense mechanism. gene encoding LL-37 in cultured epithelial cell lines were up-regulated when treated with butyrate; butyrate decreased the severity of Shigella infections in rabbit model. We could reproduce our findings from human i.e. downregulation of CAP-18 (the rabbit homologue to human LL-37) in colon epithelia after infection with Shigella flexneri. CAP-18 reappeared after treatment of the infected rabbits with sodium butyrate. Thus, the rabbit model demonstrated the proof of principal. In this study, we aim to assess the efficacy of sodium butyrate enema in reduction of clinical symptoms and / severity, reduction of inflammatory responses and induction of endogenous antibiotic activity in the rectum in adult patients with shigellosis.

DETAILED DESCRIPTION:
Study design: A double blind randomized clinical trial with subsequent follow-up.

Study Subjects: Adult male and female patients attending the Clinical Research and Service Center (CRSC) of ICDDR,B and Matlab Hospital will be screened for participation in the study.

Randomization:

According to a computer-generated randomization list, patients full filling the entry criteria will be randomized to either intervention group (Pivmecellinam plus butyrate enema) or control group (Pivmecellinam plus normal saline enema). Butyrate enema will contain 80 mmol/L of butyrate in normal saline (pH 7.2). Placebo enema will contain normal saline(pH 7.2)

Case management:

After enrollment, the patients will be admitted in the study ward of ICDDRB Dhaka and Matlab hospital. A standard clinical history and clinical examination will be performed by one of the investigators or study physician. All patients will receive Pivmecillinam, 400 mg, 8 hourly for 5 days. The intervention group will receive butyrate enema 80 ml of 80 mM sodium butyrate, 12 hourly for 72 hours while the placebo group will get 80 ml of normal saline 12 hourly for 72 hours. All patients will receive the usual hospital food three times a day (breakfast, lunch and supper). The patients will remain in the study ward for 5 days to enable identification of any relapse cases.

Procedure for butyrate enema:

Patients will be instructed to lie on a bed (cholera cot) in left lateral position. A soft rectal catheter will be introduced by a nurse/physician, through which 80 ml of butyrate solution will be instilled slowly with a 50 ml plastic syringe. Patients will be asked to retain the enema for at least ½ hour by remaining supine for 30 minutes after the administration. However, if a patient cannot retain the enema for 30 minutes, he will be given a second round of enema immediately after defecation.

Definition of clinical cure: A patient will be defined as clinically cured if on day-3, no blood or mucus is observed in the stool, there is ≤ 3 unformed stool in 24 hours and no fever (oral temperature > 37.5° C) is recorded.

Treatment failure: A patient will be considered a treatment failure on day 3 when there is any one of the following features present: > 3 unformed stool in 24 hours, presence of blood in any stool or presence of fever (oral temperature > 37.5° C).

Collection of Samples:

Patients will be requested to stay in the hospital for at least 5 days to facilitate disease monitoring and sampling. On admission day (patients will be enrolled after serological confirmation by slide agglutination test on the subsequent day i.e. day-1), stool specimens will be collected from each patient every day starting from the day of admission till 4 days after admission. Rectal biopsy samples will be collected on the day of admission and 7 days after admission from patients enrolled in Dhaka hospital only. Three mL blood will be collected after admission for measurement of C-reactive protein (CRP) that will be used as an indicator for monitoring magnitude of inflammation. 1 mL blood from patients will be collected to measure CRP in serum on the 4th day of admission.

Stool: Fresh stool samples will be collected for routine microscopic examination for parasites or cysts and as well as RBC, pus cells and macrophages. Stool samples will also be tested for measuring bacterial counts/load. In brief, 1 g of stool will be diluted in normal saline (1:10), vortex-mixed for 5 min, followed by serial dilutions of 1:10 in normal saline and plated in MacConkey agar plates. After overnight incubation at 37ºC, bacterial cfu will be counted. Fresh stool specimens will also be extracted as described earlier for measuring LL-37,human beta-defensin 1 and 3 and proinflammatory cytokines (interleukin-8 and 1beta) by ELISA method.

Rectal biopsy: Rectal biopsy samples will be obtained from patients (only in Dhaka Hospital).

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* duration of diarrhoea 0-4 days
* culture-confirmed Shigella spp (all Shigella spp) in stool on enrolment

Exclusion Criteria:

* who received antimicrobial treatment before attending the ICDDR,B hospital
* clinical symptoms of other concomitant infections (such as chronic respiratory infections, other concomitant gastrointestinal infections)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of the study is to assess the efficacy of sodium butyrate enema in adult patients with shigellosis in marked improvement in clinical, endoscopic and histological findings. | 4 years

SECONDARY OUTCOMES:
To study the effect of sodium butyrate on the induction of endogenous antibiotic peptides in the rectum in adults with shigellosis. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rubhana Raqib, Ph.D., Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (2):
- Bangladesh (2):
  - Dhaka Hospital & Matlab Hospital, Dhaka
  - ICDDR,B, Dhaka

REFERENCES:
- [Background] Raqib R, Sarker P, Bergman P, Ara G, Lindh M, Sack DA, Nasirul Islam KM, Gudmundsson GH, Andersson J, Agerberth B. Improved outcome in shigellosis associated with butyrate induction of an endogenous peptide antibiotic. Proc Natl Acad Sci U S A. 2006 Jun 13;103(24):9178-83. doi: 10.1073/pnas.0602888103. Epub 2006 Jun 1. PMID 16740661
- [Derived] Raqib R, Sarker P, Mily A, Alam NH, Arifuzzaman AS, Rekha RS, Andersson J, Gudmundsson GH, Cravioto A, Agerberth B. Efficacy of sodium butyrate adjunct therapy in shigellosis: a randomized, double-blind, placebo-controlled clinical trial. BMC Infect Dis. 2012 May 10;12:111. doi: 10.1186/1471-2334-12-111. PMID 22574737